CLINICAL TRIAL: NCT06153147
Title: KIdney aNd blooD prESsure ouTcomes in Childhood Cancer Survivors (CCS): Prospective Study
Brief Title: KIdney aNd blooD prESsure ouTcomes in Childhood Cancer Survivors (CCS)
Acronym: KINDEST-CCS
Status: Recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Michael Zappitelli, Staff Nephrologist and Senior Scientist, The Hospital for Sick Children
Other Study IDs: OCREB 4177
Record Dates: First submitted 2022-11-04; First posted 2023-12-01 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Childhood Cancer; Chronic Kidney Diseases; Hypertension; Acute Kidney Injury; Nephrotoxicity
MeSH Terms: conditions — Neoplasms; Renal Insufficiency, Chronic; Hypertension; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 5 milliliter (mL) of whole blood using Serum Separation Tubes (SST) 30 milliliter (mL) of urine 24 hour and first morning urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Late effects after nephrotoxic chemotherapies.: 3 and 5 year kidney and blood pressure effects after cancer therapy.

SUMMARY:
Background: Childhood cancer survivors (CCS) are at elevated risk of chronic health conditions. Chemotherapies can cause recurrent acute kidney injury which may progress to kidney fibrosis, chronic kidney disease (CKD) or hypertension (HTN). CCS surviving to adulthood are at ≥3 times the risk (vs. non-CCS) for CKD, HTN and lower quality of life. However, the timing of CKD and HTN onset in CCS completing cancer therapy in childhood remains unclear.

Guidelines provide recommendations on managing post-cancer therapy effects in CCS, but they lack specificity on kidney testing content, frequency and complications. This discord is largely due to knowledge gaps on which CCS develop CKD or HTN after cancer therapy, when outcomes occur and their severity. Existing work has shown in select patients, CKD and HTN in CCS likely begins in the first 5 years post-cancer therapy and that the burden is significant. With robust data on CKD and HTN, international CCS follow-up guidelines can be optimized to include detailed and actionable recommendations on kidney and blood pressure monitoring and treatment.

DETAILED DESCRIPTION:
Significant improvements in childhood cancer survival rates have come at the cost of an increase in chronic health conditions. Childhood cancer survivors (CCS) often experience chronic kidney disease (CKD) and hypertension (HTN), yet data on the onset and severity of these diseases in the primary years after childhood cancer therapy is unclear. Both CKD and HTN are major treatable cardiovascular risk factors, and the knowledge gap in the first 5 years after therapy impedes the creation of evidence-based guidelines and early intervention plans.

Currently, the Children's Oncology Group international guidelines, which are used to identify and manage therapy effects in CCS, lack information on CKD testing and appropriate measures. With appropriate treatment, CKD and HTN complications are treatable.

In 500 CCS at high risk for blood pressure (BP) and late kidney effects due to cancer therapy, we will determine the prevalence of HTN and CKD at 3 and 5 years after cancer therapy, and the extent to which eGFR, albuminuria and BP worsen from 3 to 5 years after therapy. In addition, we will assess whether acute kidney injury during cancer therapy and cardiometabolic risk factors are associated with these outcomes.

Based on the evidence from the study, we hope to improve current CCS kidney and BP guidelines to advise on appropriate treatments and measures for HTN and CKD. As CCS are vulnerable to cardiovascular disease, addressing CKD and HTN complications will improve their overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 3 years ± 6 months after therapy for first cancer
* Received high-risk therapy for first cancer, as defined by the Canadian Oncology Group (COG) as alkylating agents; platinums; abdominal or total body radiation; high dose methotrexate; stem cell transplant; nephrectomy; or other therapy which may be known to possibly cause late kidney and/or BP effects.

Exclusion Criteria:

* Pre-cancer severe CKD and/or previous kidney transplant
* >19 years old at 3 years after cancer therapy completion

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Observational cohort study of CCS at 5 Ontario child cancer centres
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2029-10-25 (Estimated); Study Completion 2039-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Chronic Kidney Disease (CKD) based on eGFR (using an equation) at 3 years post cancer therapy | 3 years +/- 6 months after cancer therapy end
  CKD: Per Kidney Disease Improving Global Outcomes (KDIGO) guidelines
Prevalence of Chronic Kidney Disease (CKD) based on eGFR (using an equation) at 5 years post cancer therapy | 5 years +/- 6 months after cancer therapy end
  CKD: Per Kidney Disease Improving Global Outcomes (KDIGO) guidelines
Prevalence of Hypertension (HTN) from office blood pressure (vis blood pressure machine) at 3 years post cancer therapy | 3 years +/- 6 months after cancer therapy end
  Defined by 2017 American Academy of Pediatrics (AAP) guidelines
Prevalence of Hypertension (HTN) using Ambulatory Blood Pressure Measurement (ABPM) at 5 years post cancer therapy | 5 years +/- 6 months after cancer therapy end
  The presence of either ambulatory hypertension or masked hypertension
Change in markers of kidney health (eGFR)(using an equation) between 3 and 5 years post cancer therapy | Change from 3 to 5 years in eGFR
  Change in eGFR in milliliter (mL) /min/1.73m2
Change in markers of kidney health (Albuminuria) (using lab values) between 3 and 5 years post cancer therapy | Change from 3 to 5 years in Albuminuria
  Change in albuminuria in mg/g
Change in markers of kidney health (Proteinuria) (using Lab values) between 3 and 5 years post cancer therapy | Change from 3 to 5 years in Proteinuria
  Change in proteinuria in mg/mmol
Change in markers of cardiovascular health (using blood tests) between 3 and 5 years post cancer therapy | Change from 3 to 5 years
  Change in BP percentile as per 2017 American Academy of Pediatrics (AAP) guidelines

SECONDARY OUTCOMES:
Impact of Acute Kidney Injury (AKI) and Cardiometabolic risk factors (using blood work) at baseline on CKD outcomes | At baseline for independent factors on CKD outcomes at 3 and 5 years
  CKD: Per Kidney Disease Improving Global Outcomes (KDIGO) guidelines

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital For Sick Children, Toronto, Ontario, Canada